CLINICAL TRIAL: NCT04215887
Title: Development of the "BreathEasy": a Non-contact, Hand-held Device for Measurement of Respiratory Rate (CPRM)
Brief Title: Noncontact, Handheld Device for Measurement of Respiratory Rate
Acronym: Breatheasy
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: SCH/13/018
Record Dates: First submitted 2016-04-01; First posted 2020-01-02 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2019-12

CONDITIONS: Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Sleep unit: Children admitted to sleep unit for sleep study
  Interventions: Device: Contactless Portable Respiratory rate Monitor
- School: Healthy children in school
  Interventions: Device: Contactless Portable Respiratory rate Monitor
- Emergency department: Children seen in triage in emergency department at SCH
  Interventions: Device: Contactless Portable Respiratory rate Monitor
- General practice: Adults or children attending general practice
  Interventions: Device: Contactless Portable Respiratory rate Monitor
- Ambulance: Adults or children in rapid response vehicle
  Interventions: Device: Contactless Portable Respiratory rate Monitor

INTERVENTIONS:
Device: Contactless Portable Respiratory rate Monitor — Novel hand-held respiratory rate monitor
  Other Names: "Breatheasy"

SUMMARY:
In the emergency department, a sick child is usually seen first by a nurse. Their job is to quickly assess how sick the child is and what immediate care is needed. The nurse will usually use electronic devices to check vital signs, such as body temperature, pulse rate and blood oxygen levels. However, the nurse normally has to manually count the respiration rate (this is the number of breaths taken each minute) because there is no suitable device which can do this automatically. Knowing the respiration rate is very important because if it is not normal, the nurse knows that the child may be seriously ill. Counting the respiration rate of sick children can be difficult and takes up a lot of time, especially if the child is upset, crying or moving about. To overcome this problem we are developing a device that automatically measures respiration rate in children. It works by directly sensing the air coming from the nose or the mouth when held at a small distance (about 30 cm) from the face. So far, the device has been shown to work in a research laboratory at Sheffield Hallam University. The aim is to develop it into a handheld, userfriendly device, ensuring that it complies with strict safety regulations. This application is to carry out an evaluation of our new device against its gold standard, on adult volunteers and on children attending Sheffield Children's Hospital for sleep studies as part of their clinical care. In the future, when nurses use the device they will easily be able to measure each child's respiration rate so that the most seriously ill children will be identified earlier and get correct treatment more quickly. This will ensure that the right children get admitted to intensive care units sooner and, in some cases, child deaths will be prevented.

ELIGIBILITY:
Inclusion Criteria:

* any person requiring and able to perform a respiratory rate measurement

Exclusion Criteria:

* people assessed as too unwell to participate by clinical team
* people for whom English is not first language as no interpreting service included in budget

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults or children requiring a respiratory rate measurement
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the experimental technique and the gold standard (contact based thermistor system). | Through study completion (less than 1 hour)
  Correlation between device respiratory rate measurement of and measurement using respiratory impedance plethysmography will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Elphick, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom